CLINICAL TRIAL: NCT02790528
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study of Statin Therapy In Patients With Vasospastic Angina
Brief Title: Statin Therapy In Patients With Vasospastic Angina
Acronym: STAVA
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding issue
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, professor of medicine, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AMCCV2016-11
Record Dates: First submitted 2016-05-26; First posted 2016-06-06 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Angina Pectoris, Variant; Statins, HMG-CoA
Keywords: statin; vasospastic angina
MeSH Terms: conditions — Angina Pectoris, Variant | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atorvastatin (Experimental): 20mg QD
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atorvastatin — 20mg QD
  Arms: Atorvastatin
Drug: Placebo — Placebo drug will be administered.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate whether statin is effective in the treatment of vasospastic angina.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 and more
* Vasospastic angina
* LDL less than 160mg/dl
* Written consent

Exclusion Criteria:

* Coronary artery stenosis more than 50% or ischemic coronary disease
* History of percutaneous coronary intervention
* Cerebrovascular diseases or peripheral
* Dyslipidemia required statin therapy
* Heart failure, arrhythmogenic right ventricular dysplasia, hypertrophic cardiomyopathy, akinesia or aneurysm on left ventricular wall, anomaly of coronary artery
* NYHA III and IV
* Arrhythmia
* Primary cardiac electrical diseases
* Cardiac pacemaker or implantable defibrillator
* Pregnancy or breast feeding
* Life expectancy less than 2 years

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The Composite Event of all-cause death, myocardial infarction, angina-related hospitalization | 3 years
  The number of events with the first occurrence of a composite event(all-cause death, myocardial infarction, angina-related hospitalization)

SECONDARY OUTCOMES:
all-cause death | 3 years
cardiac death | 3 years
cardiac arrest | 3 years
myocardial infarction | 3 years
angina-related hospitalization | 3 years
Composite event of death or myocardial infarction | 3 years
Composite event of cardiac death or myocardial infarction | 3 years
statin-related complications | 3 years
  event rate of statin-related complications

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: No
This is not a publicly funded trial.